CLINICAL TRIAL: NCT04646733
Title: Effect of a Low-carbohydrate, High-protein Ketogenic Diet on Weight and Body Composition: a Randomized Controlled Study
Brief Title: Effect of a Low-carbohydrate, High-protein Energy-restricted Diet on Weight and Body Composition Using DXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erik Ramirez Lopez (Other)
Responsible Party: Sponsor-Investigator, Erik Ramirez Lopez, Research Professor, Universidad Autonoma de Nuevo Leon
Organization: Universidad Autonoma de Nuevo Leon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: erik2020DUKAN; REPRIN-FOD-76 (Other: Assigned by the Faculty of Sports Organization)
Record Dates: First submitted 2020-11-13; First posted 2020-11-30 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Weight Loss; Body Composition
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical study. Subjects are assigned to one of two groups: the intervention group (group A or high protein diet or HPD) and the group without high protein diet or NHPD. The assignment is done with the use of MedCalc software and the option to create random groups. Both groups are treated equally except for the procedure or diet. The blind or double-blind procedure is not used in this study. Both groups are treated during the same study period. The maximum number of patients to be evaluated per day will be three. Patients are not mixed from one group or another in each evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Protein Diet Group (Experimental): The high protein diet (HPD) group is instructed to follow a low carbohydrate, high protein ketogenic diet.
  Interventions: Other: High Protein Diet Group
- No High Protein Diet Group (Active Comparator): No high protein diet (NHPD) group received an oat beverage consisted of 55 g of oats in 250 ml of water.
  Interventions: Other: No High Protein Diet Group

INTERVENTIONS:
Other: High Protein Diet Group — The high protein diet (HPD) group is instructed to follow a low carbohydrate, high protein ketogenic diet. This diet has 4 phases, two of weight loss until reaching the ideal weight (attack and cruise) and two of maintenance (consolidation and stabilization). During the first 2 phases, it allows 100 foods (28 vegetables). The first phase lasts 3-10 days and 72 high-protein, low-fat foods are allowed. In the second phase, there are alternate days between consuming the low glycemic index vegetables plus protein and the next day with just protein. The first two phases are ad libitum. Phase 3 (consolidation) aims to avoid rebound and begins the introduction of complex carbohydrates and legumes in individual servings. In phase 4 (stabilization), the subject returns to a free diet. However, three basic rules are introduced: protein one day a week, the exercise of at least 20 min/day (optional) and consumption of 3 tablespoons of oat bran/day.
  Arms: High Protein Diet Group
Other: No High Protein Diet Group — No high protein diet (NHPD) group received an oat beverage consisted of 55 g of oats in 250 ml of water. Beverage contained 1.6 g of betaG per portion according to FDA recommendations corresponding to 50 % of betaG required per day. Weekly bags containing oat mixture were provided on day 0 and in the third week of the trial. No additional instructions about diet, exercise program or pharmacological treatment was implemented.
  Arms: No High Protein Diet Group

SUMMARY:
People often choose certain diets to lose weight or to change their habits or lifestyle. The Dukan diet was created in the '70s and took on importance in the last decade. It is a 4 phase diet similar to the Atkins diet. However, this diet is aggressive in its first phase because it suppresses carbohydrates, the main source of external energy being saturated low-fat protein. Studies of this diet are scarce and have been limited to describing the contribution of micronutrients. In nutritional practice, it is often assumed that a popular high-protein or low-calorie ketogenic diet could cause rapid or unfavourable changes in a patient's weight and body composition. However, the effect of these diets in the short or long term on weight and on body fat, muscle mass and other components is not clear. This means that body composition has not been the main objective when analyzing the effect of a popular diet. For this reason, the meta-analyzes focus on weight change and the absence of body composition data is a limitation of the selected studies. Changes in body composition due to a popular diet should be evaluated with techniques such as DXA. The aim of this study is to analyze the effect of a low-carbohydrate, high-protein diet with energy restriction on weight and body composition using DXA. For this, a randomized controlled study will be used where a group will receive the diet protocol. The control group will have a normal diet, and only one oatmeal drink will be added (55 g of oats in 250 ml of water). The drink will contain 1.6 g of BetaG per serving according to FDA recommendations that correspond to the 50% BetaG required per day.

DETAILED DESCRIPTION:
The patients (n = 60) are invited through posters and social networks to recruit a group of 40 overweight subjects (20% above their ideal weight). The protocol is explained in detail to each one, and the patient and two witnesses sign the informed consent. Subjects are assigned to one of two groups: group A: high protein diet (HPD) and group B: non-high protein diet (NHPD). The NHPD is designed according to Mexican nutrition guidelines according to sex and age.

The main anthropometric and biochemical measurements and diet monitoring are performed in the body composition laboratory of the Faculty of Sports Organization (FOD). Four technicians (nutritionists) are in charge of taking the measurements and recording the data. The principal investigators review the quality of the information and the correct completion of the records. Each file will be assigned an identification number. Other nutritionists (graduate students) will be in charge of auditing the information according to the protocol guidelines. Principal Investigators will resolve any discrepancies between technicians and graduate students to ensure data recording, deletion, or reevaluation.

Each patient is asked for a prior medical examination before entering the study. The data from the external medical practitioner are compared with those provided by the patient for the present study.

The main anthropometric variables are measured with the international ISAK methodology. The DXA equipment is calibrated daily, and the result is analyzed and analyzed by a researcher who evaluates whether the measurement is reliable.

The data is recorded in printed formats that are immediately scanned to maintain readability. Later, they are recorded in an Excel sheet with the patient's identification number. In each measurement session, the database is analyzed for abnormal, extreme or unlikely data. Two independent researchers are responsible for reviewing the database every day.

Each patient is cared for by a nutrition student who accompanies him in the basic needs, clothing and transfers to the measurement equipment. At the end of the evaluation, patients receive a complimentary meal and free transportation home.

Patients are monitored through WhatsApp to verify the presence of adverse events with the diet. Also, for any questions with the procedures. All procedures are recorded in paper and electronic form. In addition, they are given an additional number in case of medical emergency or consultation with a nutritionist.

The sample size will be limited in the first stage to 30 patients. Measurements and preliminary analysis will be obtained at 0, day four and day fifteen. The last two measurements will be taken on day 42 and until the subjects reach their ideal body weight.

In the case of missing data or defective quality record, subjects will be removed.

Regarding the statistical analysis, multiple linear regression will be used, where the groups and measurements will be compared on the different measurement days. As covariates, covariates will be incorporated as initial values, age, sex, BMI, among others, will be adjusted. Descriptive statistics will be added.

ELIGIBILITY:
Inclusion Criteria:

* individuals between the ages of 20 and 30
* who were not currently consuming any drugs or were on diet or exercise treatment.
* patients must have 120% or more of the ideal weight until a BMI of 35.

Exclusion Criteria:

* with no cardiovascular disease, kidney, intestinal or liver disease.
* cholesterol (≥ 200 mg/dL)
* high triglycerides (≥ 150mg/dL)
* glucose (≥ 126mg /dL)

Ages: 20 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-05-09 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Body fat | Baseline to three months.
  Body fat measurements by DXA
Lean mass | Baseline to three months
  Lean mass measurements by DXA
Weight lost | Baseline to three months
  Weight lost through the various phases

SECONDARY OUTCOMES:
Body water | Baseline to three months
  Body water changes measured by bioelectrical impedance
Resting energy expenditure | Baseline to three months
  Energy expenditure measure by calorimetry.
Caloric and macronutrient intake | Baseline to three months
  Energy and macronutrient distribution intake. To estimate the nutrient intake is used as a weighted dietary record. Each individual weighs the items on a scale before and after consumption by three consecutive days. Scales has a precision of 1 g. The persons record all the food and beverages consumed, including ingredients, preparation method, and quantity of the food consumed and not consumed. We proportionate all the instruction and description for the individual before assigning the task to record. This procedure ensures the accuracy and reliability of the information provided. Records are processed with the software DietOrganizer (R) to obtain caloric and macronutrient intake.
Serum fasting triglycerides | Baseline to three months
  Serum fasting triglicerides are taken after 9 to 12 h, milligrams per deciliter (mg/dL).
Serum fasting glucose | Baseline to three months
  Serum fasting glucose is taken after 9 to 12 h, milligrams per deciliter (mg/dL).
Serum fasting total cholesterol | Baseline to three months
  Serum total cholesterol is taken after 9 to 12 h, milligrams per deciliter (mg/dL).
Serum fasting HDL cholesterol | Baseline to three months
  Serum total cholesterol is taken after 9 to 12 h, milligrams per deciliter (mg/dL).
Serum fasting albumin | Baseline to three months
  Serum total cholesterol is taken after 9 to 12 h, grams per deciliter (g/dL).
Serum fasting total protein | Baseline to three months
  Serum total cholesterol is taken after 9 to 12 h, grams per deciliter (g/dL).
Serum fasting total hemoglobin | Baseline to three months
  Serum total cholesterol is taken after 9 to 12 h, grams per deciliter (g/dL).
hand strenght with a dynamometer | Baseline to three months
  Hand strength is measured with a standardized protocol using a chair. A digital dynamometer is employed, and units are expressed as kg.
triceps skinfold with a plicometer | Baseline to three months
  triceps skinfold is measured with a plicometer and the units are expresed as mm
waist perimeter | Baseline to three months
  waist perimeter is measured with a measuring tape and units are expresed as cm
mid-arm perimeter | Baseline to three months
  mid arm perimeter is measured with a measuring tape and units are expresed as cm

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Organización Deportiva, FOD, Universidad Autónoma de Nuevo León, Monterrey, N.L., Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anton SD, Hida A, Heekin K, Sowalsky K, Karabetian C, Mutchie H, Leeuwenburgh C, Manini TM, Barnett TE. Effects of Popular Diets without Specific Calorie Targets on Weight Loss Outcomes: Systematic Review of Findings from Clinical Trials. Nutrients. 2017 Jul 31;9(8):822. doi: 10.3390/nu9080822. PMID 28758964
- [Background] Atallah R, Filion KB, Wakil SM, Genest J, Joseph L, Poirier P, Rinfret S, Schiffrin EL, Eisenberg MJ. Long-term effects of 4 popular diets on weight loss and cardiovascular risk factors: a systematic review of randomized controlled trials. Circ Cardiovasc Qual Outcomes. 2014 Nov;7(6):815-27. doi: 10.1161/CIRCOUTCOMES.113.000723. Epub 2014 Nov 11. PMID 25387778
- [Background] Seid H, Rosenbaum M. Low Carbohydrate and Low-Fat Diets: What We Don't Know and Why we Should Know It. Nutrients. 2019 Nov 12;11(11):2749. doi: 10.3390/nu11112749. PMID 31726791